CLINICAL TRIAL: NCT05628285
Title: Evaluation of a Sound Processor for a Transcutaneous System
Brief Title: Evaluation of a Hearing Device for Transmitting Sound to the Inner Ear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC114
Record Dates: First submitted 2022-11-08; First posted 2022-11-28 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Conductive Hearing Loss; Mixed Hearing Loss
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sentio 1 sound processor (Experimental): The sound processor picks up the sound and transfer it to the implant that convert the sound to vibrations that are transmitted to the inner ear.
  Interventions: Device: Sentio 1

INTERVENTIONS:
Device: Sentio 1 — Sound processor

SUMMARY:
A single center study evaluating the performance of an externally worn sound processor for a transcutaneous bone anchored hearing system using audiological outcomes measures such as aided thresholds and self-evaluation questionnaires.

DETAILED DESCRIPTION:
Bone conduction hearing systems use the body's natural ability to transfer sound through bone conduction. The sound processor picks up sound and converts it into vibrations that are transferred through the skull bone to the inner ear (cochlea). Thus, for patients with conductive or mixed hearing losses, patients with lasting hearing loss following a middle ear disease or malformations (such as microtia), the vibrations are bypassing the conductive problem in the ear canal or middle ear. Bone conduction devices currently on the market are divided into three types; transcutaneous direct drive, percutaneous (skin penetrating) direct drive and transcutaneous skin drive bone conduction devices. This evaluation focus on a sound processor used for a transcutaneous system.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Adult subjects (18 years or older)
3. Subjects implanted with an I1 implant
4. Fluent in Swedish

Exclusion Criteria:

1. Subjects who do not have the ability or are un-willing to follow investigational procedures/requirements, e.g., to complete questionnaires, according to investigator's discretion.
2. Subject deemed unsuitable for any medical or other reason as judged by PI or medical responsible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2024-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Charlotte Persson, Principal Investigator — Habilitation & Health, Hearing organization Södra Gubberogatan 6, 416 63 Göteborg, Sweden
Locations (1):
- Habilitation & Health, Hearing organization, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Ears
Period: Overall Study
Arm/Group | Sentio 1 Sound Processor
Started | 11; 11 Ears
Completed (Study is still ongoing. 10 subjects have completed the primary endpoint visit (1 month follow-up) and are still active in the study.) | 10; 10 Ears
Not Completed | 1; 1 Ears
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sentio 1 Sound Processor
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 51 [27 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Improvement of Hearing With the Sentio1 (PTA4)
Description: Functional gain with Sentio 1, i.e., the difference in dB between unaided and aided sound field thresholds, calculated on average for frequencies 500, 1000, 2000 and 4000 Hz (PTA4).
  In detail, for each patient, sound field thresholds are measured at the frequencies 500, 1000, 2000 and 4000 Hz for which a mean value is calculated and denoted as PTA4.
  The primary outcome measure is functional gain which is the difference in PTA4 measured unaided (without sound processor) versus aided condition (with sound processor).
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: dB
Units Other Than Participants: Ears
Groups:
- Functional Gain PTA4 (Sentio 1 Sound Processor): The sound processor picks up the sound and transfer it to the implant that convert the sound to vibrations that are transmitted to the inner ear.
  Sentio 1: Sound processor
Arm/Group | Functional Gain PTA4 (Sentio 1 Sound Processor)
Number analyzed (Participants) | 10
Number analyzed (Ears) | 10
dB | 32.5 (6.8)

2. Secondary Outcome: To Assess the Improvement of Hearing With the Sentio1
Description: Functional gain with Sentio 1, i.e., the difference in dB between unaided (without sound processor) and aided (with sound processor on) sound field thresholds, for all measured frequencies.
  In detail, for each patient, sound field thresholds are measured at the frequencies 250, 500, 1000, 2000, 3000, 4000, 6000 and 8000 Hz, with and without the sound processor on.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: dB
Units Other Than Participants: Ears
Groups:
- Functional Gain (All Frequencies) (Sentio 1 Sound Processor): The sound processor picks up the sound and transfer it to the implant that convert the sound to vibrations that are transmitted to the inner ear.
  Sentio 1: Sound processor
Arm/Group | Functional Gain (All Frequencies) (Sentio 1 Sound Processor)
Number analyzed (Participants) | 10
Number analyzed (Ears) | 10
dB
  250Hz | 18.5 (11.6)
  500Hz | 29.5 (12.1)
  1000Hz | 35.0 (6.2)
  2000Hz | 33.5 (10.3)
  3000Hz | 35.0 (13.1)
  4000Hz | 32.0 (8.9)
  6000Hz | 23.5 (9.1)
  8000Hz | 17.8 (12.9)

3. Secondary Outcome: Subjective Evaluation of Sound Processor Performance.
Description: Sentio 1 compared to previous sound processor.
  1. Average SSQ12 scores with Sentio 1 for each question, sub-scales and in total.
  2. Average SSQ12 scores with current sound processor for each question, sub-scales and in total.
  3. Difference in SSQ12 scores between Sentio 1 and current sound processor for each question, sub-scales and in total.
  Measured by the Speech, Spatial and Quality (SSQ) scale from 0-10 where 0 represents "Not at all" and 10 represents "Perfect". Higher scores mean a better outcome. For each of the scales the item outcomes are averaged. Fot the total score all items are averaged
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Ears
Groups:
- Previous Sound Processor: Measurement at Visit 1 with the patient's own sound processor
- Sentio 1 Sound Processor: Measurement at Visit 2 with the Sentio 1 sound processor
- Difference Between Visit 2 (Sentio 1) and Visit 1 (Previous Device): Visit 2 (Sentio 1) - Visit 1 (previous device)
Arm/Group | Previous Sound Processor | Sentio 1 Sound Processor | Difference Between Visit 2 (Sentio 1) and Visit 1 (Previous Device)
Number analyzed (Participants) | 11 | 10 | 10
Number analyzed (Ears) | 11 | 10 | 10
score on a scale
  SSQ Speech | 5.58 (2.32) | 6.07 (2.67) | 0.579 (1.537)
  SSQ Spatial | 4.34 (3.02) | 4.68 (2.90) | 0.353 (1.590)
  SSQ Quality | 6.21 (2.12) | 6.22 (1.70) | 0.154 (0.920)
  SSQ Total | 5.47 (2.18) | 5.78 (2.26) | 0.402 (0.937)

4. Secondary Outcome: Subjective Sound Processor Preference
Description: Percentage (%) of subjects who prefer the Sentio 1 over current sound processor
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Sentio 1 Sound Processor
Number analyzed (Participants) | 10
Participants | 7

5. Secondary Outcome: To Assess the Degree to Which Sentio 1 Compensates for the BC Hearing Loss
Description: 1. Effective gain defined as the difference in dB between aided sound field thresholds with Sentio 1 and unmasked BC thresholds on the aided ear(s). The effective gain is calculated for all measured frequencies.
  2. Effective gain with Sentio 1, see definition above, calculated in average for frequencies 500, 1000, 2000 and 4000 Hz (PTA4).
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: dB
Groups:
- Effective Gain (Sentio 1): Aided threshold - Unmasked BC threshold
Arm/Group | Effective Gain (Sentio 1)
Number analyzed (Participants) | 10
dB
  500Hz | 20.5 (13.6)
  1000Hz | 11.0 (7.4)
  2000Hz | 1.50 (10.01)
  3000Hz | 12.5 (9.2)
  4000Hz | 14.5 (9.0)
  PTA4 | 11.9 (7.7)

6. Secondary Outcome: To Assess the Difference Between BC In-situ Thresholds Measured With Sentio 1 and Conventional Unmasked BC Audiometry.
Description: Difference in dB between Sentio 1 BC in situ thresholds and BC thresholds measured with conventional unmasked BC audiometry for the frequencies 500, 1000, 2000, 3000 and 4000 Hz.
  The BC in-situ threshold is a measure of the inner ear functionality with the device. This should correspond to the unmasked BC thresholds measured with conventional audiometry. The difference was calculated as the threshold value measured with Sentio 1 minus the threshold value measured with conventional audiometry. Negative values indicate that the thresholds measured with Sentio 1 were lower (better) compared to those measured with conventional audiometry. Conversely, positive values indicate that the thresholds measured with Sentio 1 were higher (worse) compared to conventional audiometry. It's expected that two measurements should be comparable to each with a difference of maximum +/-5 dB.
Time Frame: 1 month
Measure: Mean (Standard Error); unit: dB
Units Other Than Participants: Ears
Groups:
- Difference Between BC In-situ Thresholds and Conventional Unmasked BC Audiometry: The sound processor picks up the sound and transfer it to the implant that convert the sound to vibrations that are transmitted to the inner ear.
  Sentio 1: Sound processor
Arm/Group | Difference Between BC In-situ Thresholds and Conventional Unmasked BC Audiometry
Number analyzed (Participants) | 11
Number analyzed (Ears) | 11
dB
  500Hz | -4.7 (11.5)
  1000Hz | -3.4 (9.0)
  2000Hz | -6.7 (7.9)
  3000Hz | 8.2 (8.4)
  4000Hz | 9.9 (9.2)

7. Secondary Outcome: Assess Safety With the Sentio 1 Sound Processor
Description: Tabulation of AEs occurred throughout the investigation and percentage of individuals with reported AEs.
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From enrollment up to 24 months
Arm/Group | Sentio 1 Sound Processor
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT05628285/Prot_SAP_000.pdf